CLINICAL TRIAL: NCT02755194
Title: "Drugs in Lactation" Analysis Consortium (DLAC)
Brief Title: "Drugs in Lactation" Analysis Consortium
Acronym: DLAC
Status: Terminated | Type: Observational
Why Stopped: This infrastructure project has been taken over by another study.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Shinya Ito, Division Head, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000036538
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Lactation
Keywords: pharmacokinetics; Drug-in-milk; breastfeeding; drug safety; population pharmacokinetics
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Breast milk samples are collected at different time-points before and after taking the medication.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breastfeeding women on the study medications: The study population consists of lactating/breastfeeding women over the age of 18, who are able to communicate in English and are taking one or more of the study drugs (Infliximab, Adalimumab, Golimumab, Certolizumab, Etanercept, Methotrexate, Ezetimibe, Bupropion, Citalopram, Venlafaxine)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. The exposure of interest includes taking specific prescribed medications during breastfeeding.

SUMMARY:
Some medications taken by the breastfeeding women are excreted into milk, posing a potential risk of toxicity to the infant. The first line of evidence required for toxicity risk assessment is prediction of drug levels in milk. However, pharmacokinetic (PK) information of drug excretion into milk is largely lacking, or limited to data from case reports. This makes it difficult to provide population-level prediction of drug levels in milk. The lack of data on this topic jeopardizes not only maternal adherence to drug therapy during breastfeeding but also establishment of breastfeeding, even if the drug is considered safe during nursing. Clearly, this clinical problem in drug safety is an important women's health issue, affecting both mother and infant. "Drugs in Lactation" Analysis Consortium (DLAC) is a "drug-in-milk" monitoring network, which is designed as a platform for efficient collection of patient milk samples in a real world setting to generate population predictions of drug excretion levels into human milk.

DETAILED DESCRIPTION:
OVERARCHING GOAL OF DLAC:

To establish a post-marketing "drug-in-milk" monitoring system for nursing women who are prescribed and using medications. Drugs in Lactation Analysis Consortium (DLAC) will provide risk assessment data and tools for toxicity detection in the form of population estimates and variations of drug levels in mother's milk and infant plasma for several common medications in a real world setting.

SPECIFIC OBJECTIVES:

* To generate data on drug levels in breast milk
* To develop a population pharmacokinetic model describing drug levels in milk
* To simulate/predict drug levels in milk in a population, based on the pop PK model
* To develop a physiologically-based pharmacokinetic (PBPK) model describing drug levels in infant serum
* To screen the breastfed infants of mothers on the study drugs for general health condition (medical issues, developmental milestones)

SCOPE AND RATIONALE:

Information on the extent of drug excretion into mother's milk is lacking, mainly due to the following two reasons: 1) nursing women are excluded from drug trials; 2) ethical and practical difficulties in conducting intensive-sampling PK studies in the breastfeeding mothers. Even if data exist, they are based on small numbers of patients, and it is difficult to translate the information into population estimates of drug levels in milk. DLAC is developed as a novel drug safety network using population PK (popPK) modeling approach, which allows population-level PK parameter estimation, modeling and simulation based on a scheme of sparse sampling per individual, systematically collected from a large number of nursing women on medication in real world setting. This approach will provide population risk estimates as probability distribution of reaching certain drug level in milk and plasma. Equipped with a versatile drug analysis core and a popPK modeling and simulation unit, DLAC will be able to generate PK estimates of a population in the context of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old Taking one or more drugs of interest of the study, at steady state

Exclusion Criteria:

* Being unable to communicate in English, Colostrum phase (<1 week postpartum)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lactating women over the age of 18 who are taking one of the drugs of interest of the study
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Drug levels in breast milk | Through the study completion, an average of 4 years
  Robust parameter estimates from pop PK modelling usually require samples from >30-50 individuals. Therefore, an average of 4 years is considered as the time frame, so that the required numbers of samples for each drug can be collected for population PK analysis and modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Shinya Ito, MD, FRCPC, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No